CLINICAL TRIAL: NCT02731911
Title: Phase 4, Open-label, Non-randomized, Prospective Study of OZURDEX® in the Treatment of Diabetic Macular Oedema - The AUSSIEDEX Study
Brief Title: Study of OZURDEX® in the Treatment of Diabetic Macular Oedema (DME) in Australia - The AUSSIEDEX Study
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: CMO-AP-EYE-0438
Record Dates: First submitted 2016-03-24; First posted 2016-04-08 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Macular Oedema
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ozurdex® (dexamethasone intravitreal implant): Patients who received Ozurdex® in the treatment of Diabetic Macular Oedema per local standard of care in clinical practice.
  Interventions: Drug: dexamethasone intravitreal implant

INTERVENTIONS:
Drug: dexamethasone intravitreal implant — Ozurdex® treatment for diabetic macular oedema as per standard of care in clinical practice.

SUMMARY:
This prospective study will assess Ozurdex in the treatment of Diabetic Macular Oedema in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pseudophakic or phakic and scheduled for a cataract operation
* Macular oedema due to DME

Exclusion Criteria:

* Previous Ozurdex® treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are pseudophakic, or phakic and scheduled for a cataract operation, and with a diagnosis of Diabetic Macular Oedema in one or both eyes who are to be treated with Ozurdex® at least once as determined by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 202 (Actual)
Dates: Start 2016-04-29 (Actual); Primary Completion 2018-10-22 (Actual); Study Completion 2018-10-22 (Actual)

PRIMARY OUTCOMES:
Mean change in Best Corrected Visual Acuity (BCVA) from baseline | Baseline, Month 12
Mean change in Central Retinal Thickness (CRT) from baseline | Baseline, Month 12

SECONDARY OUTCOMES:
Percentage of patients with a BCVA improvement of 15 letters or more | Baseline, Month 12
Percentage of patients with a BCVA improvement of 10 letters or more | Baseline, Month 12
BCVA average mean from baseline in area under the curve (AUC) analysis | Baseline, Month 12
Number of Intraocular Pressure (IOP)-lowering treatments used to control IOP increase | 12 Months
Mean BCVA at each injection number | 12 Months
Mean change from baseline in BCVA at each injection number | Baseline, Month 12
Mean change in BCVA across all the study injection numbers | Baseline, 12 Months
Percentage of patients with BCVA improvement | Baseline, Month 12
Percentage of BCVA losers | Baseline, Month 12
Percentage of patients improving to 20/40 or better | Month 12
Mean number of Ozurdex injections | 12 Months
Mean interval between Ozurdex® injections | 12 Months
Change from baseline in central subfield retinal thickness by Optical Coherence Tomography (OCT) before each follow-up injection number | Baseline, Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. George Labib, Study Director — Allergan
Locations (23):
- Australia (23):
  - Retina and Macula Specialists,Hurstville, Hurtsville, New South Wales
  - Retina Associates, Liverpool, New South Wales
  - Retina and Macula Specialists, Miranda, Miranda, New South Wales
  - Eye Doctors Mona Vale, Mona Vale, New South Wales
  - Marsden Eye Clinic, Parramatta, New South Wales
  - Retina & Vitreous Centre Strathfield, Strathfield, New South Wales
  - Strathfield Retina, Strathfield, New South Wales
  - Retina & Vitreous Centre City, Sydney, New South Wales
  - Sydney Eye and Retina Clinic, Sydney, New South Wales
  - Sydney Eye Hospital/Macular Diseases Centre, Sydney, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - Terrace Eye Centre, Brisbane, Queensland
  - Caboolture Eye Surgery, Caboolture, Queensland
  - Peninsula Eye Hospital, Redcliffe, Queensland
  - The Qld Eye Institute, South Brisbane, Queensland
  - Adelaide Eye & Retina Centre, Adelaide, South Australia
  - Department of Opthalmology, Royal Adelaide Hospital, Adelaide, South Australia
  - Hobart Eye Surgeons, Hobart, Tasmania
  - Tasmanian Eye Institute, Launceston, Tasmania
  - Essendon Retina, Essendon, Victoria
  - Victoria Parade Eye Consultants, Fitzroy, Victoria
  - Vision Eye Institute, Footscry, Victoria
  - Lions Eye Institute, Nedlands, Western Australia

REFERENCES:
- [Derived] Mitchell P, Arnold J, Fraser-Bell S, Kang HK, Chang AA, Tainton J, Simonyi S. Dexamethasone intravitreal implant in diabetic macular oedema refractory to anti-vascular endothelial growth factors: the AUSSIEDEX study. BMJ Open Ophthalmol. 2023 Aug;8(1):e001224. doi: 10.1136/bmjophth-2022-001224. PMID 37541745
- [Derived] Fraser-Bell S, Kang HK, Mitchell P, Arnold JJ, Tainton J, Simonyi S. Dexamethasone intravitreal implant in treatment-naive diabetic macular oedema: findings from the prospective, multicentre, AUSSIEDEX study. Br J Ophthalmol. 2023 Jan;107(1):72-78. doi: 10.1136/bjophthalmol-2021-319070. Epub 2021 Aug 25. PMID 34433549